CLINICAL TRIAL: NCT03358979
Title: Three-dimensional Analysis of EMMPRIN on Conjunctival Epithelial Cells Surface in Severe Dry Eye Syndrome (ALTESSE)
Acronym: ALTESSE
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: EGN_2017_15
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Conjunctival Diseases; Dry Eye Syndromes
Keywords: Conjunctival Diseases; Dry Eye Syndromes; Antigens; CD147
MeSH Terms: conditions — Conjunctival Diseases; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe eye dryness
- absence of eye dryness

SUMMARY:
Modifications of cell surface markers (including EMMPRIN) were observed in conjunctival epithelial cells during dry eye syndrome ; this study aims to describe the modifications of the repartition of these cell surface markers before and after initiation of a treatment.

ELIGIBILITY:
Patients:

Inclusion criteria

* 18 years and over
* Severe eye dryness (grade 3 or 4) as defined by the International Dry Eye Work Shop (2007): Frequent symptoms, Impregnation of fluorescein at the conjunctival level, marked fluorescein staining at the corneal level, Tear Break Up Time ≤ 5 seconds (fluorescein test) Schirmer's test score without anesthesia ≤ 5mm at 5 minutes
* Patients without eye treatment or patients undergoing long-term stable eye treatment for whom a new treatment is being introduced

Exclusion criteria - Known pregnancy or breastfeeding

Control subjects:

Inclusion criteria

- 18 years and over

Exclusion criteria

* Wearer of contact lenses
* Topical ocular treatment
* Known pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe eye dryness will be compared with persons without eye dryness.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
comparison of surface area of cell markers measured on conjunctival epithelial cells, in persons with and without severe eye dryness. | baseline
  Comparison of the mean surface in patients before treatment for eye dryness versus in persons with no eye dryness. Immunofluorescence analysed in confocal microscopy on conjunctival impression cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Eric GABISON, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A de Rothschild, Paris, France